CLINICAL TRIAL: NCT06336226
Title: Brachio Basilic Arterio Venous Fistula One Stage Versus Two Stage as a Hemodialysis Access
Brief Title: Brachio Basilic Arterio Venous Fistula One Stage vs Two Stage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelrasheed Mohamed Abdelrasheed, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BB AVF one stage vs two stage
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Arterio-venous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One stage group (Active Comparator): The one-stage operation was performed under regional anesthesia. A 5-cm incision at the ante cubital fossa identifies the basilic vein. The incision was extended proximally, and the underlying deep fascia was opened. The basilic vein was mobilized up to its junction with the brachial vein. The median cutaneous nerve of the forearm was carefully dissected and preserved. After side branches were ligated, the basilic vein was tunnelled subcutaneously, with a Roberts' forceps maintaining its axial orientation.An end-to-side arteriovenous anastomosisto the brachial artery was performed
  Interventions: Procedure: Brachio basilic arterio venous fistula one stage versus two stage
- two stage group (Active Comparator): he first stage of the two-stage procedure was performed under local anesthesia by formation of the arteriovenous anastomosis with minimal disturbance of the basilic vein. After 4 to 6 weeks, a flow assessment of the AVF by duplex scanning was made to determine if revision of the anastomosis was necessary at the second stage. The second stage was performed under regional anesthesia. The entire length of the basilic vein was mobilized, a"subcutaneous flap" was created, and the vein was positioned anterolaterally. Usually, a further 2 weeks was required before the AVF can be used
  Interventions: Procedure: Brachio basilic arterio venous fistula one stage versus two stage

INTERVENTIONS:
Procedure: Brachio basilic arterio venous fistula one stage versus two stage — Comparative study between one stage brachio basilic arterio venous fistula versus two stage

SUMMARY:
The aim of this work was to compare primary failure rates and the primary functional patency of one-stage vs two stage brachiobasilic fistulas to compare the two surgical techniques .

DETAILED DESCRIPTION:
In the last two decades, there have been concerted efforts by the National Kidney Foundation Dialysis Outcomes Quality Initiative (NKF-DOQI), and the Fistula First Breakthrough Initiative to decrease the use of prosthetic grafts and increase autogenous (native) arteriovenous fistula(AVF) creation for hemodialysis access. When considering vascular access for hemodialysis on the basis of patency, resistance to infection,and associated complications, Native AVF should be selected as the first choice whenever possible. If the cephalic vein in the upper arm is unusable for AVF construction, the basilic vein can be superficialized and anastomosed to the brachial artery at the elbow to form a brachiobasilic arteriovenous fistula (BB)AVF .

If a BB AVF is to be constructed,duplex ultrasound should be used to check the path and size of the basilic vein. It is also important to determine if an adequate length can be mobilized .

The BB fistulae can be formed in one stage or two stages. To date, limited and conflicting data exist regarding primary failure and the patency rates of one-stage and two-stage procedures. Each procedure has advantages and disadvantages Both one-stage and two-stage procedures have their advantages and disadvantages.

Which procedure results in improved outcomes remains unclear. However, the basic principle is to superficialize the basilic vein and make it amenable to needle puncture.

ELIGIBILITY:
Inclusion Criteria:

* All patients with end-stage renal disease who had their BBAVFs created either by the one-stage or two- stage technique.
* Patients with brachial artery diameter more than 3 . mm by duplex ultrasound (DUS).
* Patients with triphasic brachial artery by DUS.
* Patients with basilic vein diameter more than 3 mm by DUS.
* Patients who were able to give informed consent.
* Requirements for intervention agreement between the patient and the surgeon.
* Availability of patients for all follow-up visits.

Exclusion Criteria:

* Patients who already had a suitable cephalic vein for arteriovenous fistula creation.
* Patients whose brachial artery diameter was less than 3 mm by DUS.
* Patients with brachial artery disease proved by DUS.
* Patients whose basilic vein diameter was less than mm by DUS.
* Patients with ischemic cardiomyopathy.
* Patients with central venous stenosis or occlusion evidenced by duplex scanning.
* Patients with flexion deformity or skin lesions at the site of the fistula or over the course of the vein.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Comparative study between one stage brachio basilic arterio venous fistula versus two stage | 1 year
  Measures were primary fistula failure rates and patency rates at specific checkpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham A Hasan, Professor, Study Chair — Assiut University; Ahmed Kh Sayed, Lecturer, Study Director — Assiut University; Wael A Abdelgawad, Lecturer, Principal Investigator — Al-Azhar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashar K, Healy DA, Elsheikh S, Browne LD, Walsh MT, Clarke-Moloney M, Burke PE, Kavanagh EG, Walsh SR. One-stage vs. two-stage brachio-basilic arteriovenous fistula for dialysis access: a systematic review and a meta-analysis. PLoS One. 2015 Mar 9;10(3):e0120154. doi: 10.1371/journal.pone.0120154. eCollection 2015. PMID 25751655
- [Background] Kakkos SK, Lampropoulos GC, Nikolakopoulos KM, Tsolakis IA, Papadoulas SI, Papachristou EC, Goumenos D, Lazarides MK. A Systematic Review and Meta-Analysis of Randomized Trials Comparing Two-Stage with One-Stage Brachio-Basilic Vein Fistulas. Vasc Specialist Int. 2018 Sep;34(3):51-60. doi: 10.5758/vsi.2018.34.3.51. Epub 2018 Sep 30. PMID 30310807